CLINICAL TRIAL: NCT00882986
Title: Role of Exercise Training and Body Weight on Cardiovascular and Metabolic Responses to a Mixed Meal Tolerance Test
Brief Title: Cardiovascular and Metabolic Responses to a Mixed Meal
Status: Completed | Type: Observational
Sponsor: John Thyfault (Other)
Responsible Party: Sponsor-Investigator, John Thyfault, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 1121717
Record Dates: First submitted 2009-04-14; First posted 2009-04-17 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Insulin Resistance
Keywords: insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Men with high fitness (above VO2max of 60)
- 2: Men with average fitness (below VO2max of 50)

SUMMARY:
The purpose is to determine whether regular endurance exercise and/or body weight influence the way our nervous and vascular systems respond during the metabolism of meals.

DETAILED DESCRIPTION:
To begin to examine this question we recruited healthy endurance-trained (high fit, HF) and normally active (average fit, AF) subjects. It is well characterized that chronic endurance training results in enhanced peripheral insulin sensitivity. Therefore, our rationale was that inclusion of two healthy subject groups, with distinct differences in insulin sensitivity, would allow us to investigate how enhanced insulin sensitivity influences insulin-mediated changes in central sympathetic outflow. Direct measurements of central sympathetic outflow to skeletal muscle (i.e., MSNA) were recorded, and a mixed meal was used as a physiological method to evoke robust and sustained increases in MSNA, which have been primarily attributed to insulin. We hypothesized that HF subjects would have a greater MSNA response, for a given plasma insulin concentration, following consumption of a mixed meal (i.e., greater central insulin sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* healthy, not currently taking any medications

Exclusion Criteria:

* unhealthy, taking medications

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young, lean, healthy men
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
insulin/glucose response to mixed meal ingestion | This study is cross-sectional. Primary and secondary measures will be assessed at a single timepoint.

SECONDARY OUTCOMES:
MSNA | This is a cross-sectional study. Primary and seconardy measures will be assessed at a single visit lasting 4-6 hours.
Blood flow | This is a cross-sectional study. Primary and seconardy measures will be assessed at a single visit lasting 4-6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States